CLINICAL TRIAL: NCT06082713
Title: Extracellular Vesicles As Non-Invasive Biomarkers for Huntington Disease Progression and Huntingtin Lowering Therapy
Brief Title: Extracellular Vesicles for HD
Status: Recruiting | Type: Observational
Sponsor: University of Central Florida (Other)
Collaborators: University of South Florida (Other)
Responsible Party: Sponsor
Other Study IDs: STUDY00004597
Record Dates: First submitted 2023-10-08; First posted 2023-10-13 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Huntington Disease
Keywords: HD; Huntington Disease; Healthy
MeSH Terms: conditions — Huntington Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Huntington Disease Carriers
- Non-Huntington Disease Carriers

SUMMARY:
The primary objective of this study is to discover blood-based biomarker of brain Huntingtin (HTT) protein using extracellular vesicles to be used in evaluating target engagement in HTT lowering clinical trials.

Secondary objectives of this study include developing more accurate biomarkers of Huntington disease (HD) progression or conversion and to develop standard practices for extracellular vesicle biomarker discovery research.

The investigators hypothesize that brain-derived extracellular vesicles (EVs) isolated from human biofluids contain biological cargo specific to their tissue of origin that could allow their use as brain biomarkers for HD. EVs are lipid bilayer-delimited particles that are naturally released from cells in the brain.

The investigators will investigate if EVs contents reflect the pathological alterations occurring with disease progression when compared with EVs isolated from biofluids of healthy non-HD persons.

ELIGIBILITY:
Inclusion Criteria:

1. 18 - 75 years of age
2. can provide informed consent
3. able to read and speak English
4. agree to comply with study procedures (including overnight fasting, blood collection and lumbar puncture); and
5. has been diagnosed with HD (HD Carriers) or not been diagnosed with HD (Non-HD Carriers).

Exclusion Criteria:

1. younger than 18 or older than 75 years old
2. known to carry an intermediate CAG repeat between 27 and 39 or a larger expansion of 60 or more CAG repeats
3. receiving nutrition through a tube
4. pregnant
5. participated in a clinical drug trial within 30 days
6. use prescribed or non-prescribed medications that are not compatible with collection of the study samples (those that may cause excessive bleeding or prevent clotting)
7. positive for HIV, hepatitis B or C
8. have a confirmed or suspected immunodeficient condition/state
9. significant medical, psychiatric, or neurological morbidity is observed by the clinic physician on the day of sample collection that might impair completion of the study procedures
10. have needle phobia, frequent headache, significant lower spinal deformity or major surgery
11. received antiplatelet or anticoagulant therapy within 14 days prior to sample collection (including but not limited to: aspirin, clopidogrel, dipyridamole, warfarin, dabigatran, rivaroxaban and apixaban)
12. have a blood clotting or bruising disorder
13. do not comply with or are unwilling to undertake any of the study procedures

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will enroll HD carriers (HD Carriers) and non-carriers (Non-HD Carriers).
  100 participants will be enrolled. 25 from Central Florida Center for Huntington Disease at the University of Central Florida (Orlando) and 75 from Huntington's Disease Center of Excellence at the University of South Florida (Tampa).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-10-25 (Actual); Primary Completion 2031-11 (Estimated); Study Completion 2031-11 (Estimated)

PRIMARY OUTCOMES:
To discover blood-based biomarker of brain HTT protein using extracellular vesicles to be used in evaluating target engagement in HTT lowering clinical trials. | 1 year

SECONDARY OUTCOMES:
To develop more accurate biomarkers of HD progression or conversion | 8 years
to develop standard practices for extracellular vesicle biomarker discovery research | 8 years

CONTACTS AND LOCATIONS:
Overall Officials: Amber Southwell, PhD, Principal Investigator — University of Central Florida Burnett School of Biomedical Sciences
Locations (1):
- University of Central Florida, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No